CLINICAL TRIAL: NCT06197828
Title: Development and Application of Novel Biomarkers and Clinical Indicators for Early Renal Injury in Children With Sepsis
Brief Title: Novel Biomarkers for Early Renal Injury in Children With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-23-003
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury; Sepsis; Gout Flare
Keywords: pediatric, kidney injury, sepsis, gut microbiota, blood metabolome
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Upon admission, a comprehensive set of tests was conducted over a span of three consecutive days to gather essential data. These tests included blood gas analysis, urine gas analysis, routine biochemical analysis, stool analysis, and the measurement of inflammatory indicators such as CRP, IL-6, TNF-α, and PCT. Considering the regular daily monitoring of blood gas, biochemical, and urinary gas levels for critically ill patients in the ICU, no additional blood samples were drawn during this session. Instead, the routine test results were directly recorded. Parameters such as pH, PaO2, PaCO2, and the PaO2/FiO2 ratio were obtained from the blood gas analysis, while the urine gas analysis provided measurements of pH, PuCO2, and PuO2. Key indicators of renal function, such as Cr and NGAL, were also recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis-associated acute kidney injury: Between May 2021 and December 2024, patients admitted to the Pediatric Intensive Care Unit (PICU) for a duration exceeding three days were included in the study. Specifically, patients diagnosed with sepsis were selected based on the 2005 international standard for childhood sepsis, the 2012 Surviving Sepsis Campaign guidelines for pediatric sepsis, and the 2015 expert consensus on sepsis criteria for Chinese children with septic shock. The age range of the patients included in the study varied from 1 month to 16 years old.
  Interventions: Other: This study is an observational studie which have no intervention
- Patients without sepsis In ICU: patients admitted to the Pediatric Intensive Care Unit (PICU) for a duration exceeding three days and those without sepsis were included in the study.
  Interventions: Other: This study is an observational studie which have no intervention

INTERVENTIONS:
Other: This study is an observational studie which have no intervention — This study is an observational studie which have no intervention

SUMMARY:
Toxicosis often leads to multiple organ failure (MODS), with the kidney being the primary target organ due to its sensitivity to infection and ischemia. The kidney's vulnerability makes it a potential early indicator of organ failure, implying that further organ failure may occur later, thereby increasing the risk of patient mortality. Several studies conducted on sepsis patients in the Pediatric Intensive Care Unit (PICU) have revealed that 40.32% of sepsis patients experienced complications with acute kidney injury (AKI), and the case fatality rate could rise to 70% once AKI occurred. The Kidney Disease Improving Global Outcomes (KDIGO) scale is commonly used as a diagnostic criterion for AKI. However, the kidney's robust reserve function poses a challenge for early identification, diagnosis, and intervention of AKI since significant increases in creatinine levels and a sharp decrease in urine volume already indicate severe kidney damage. This situation calls for the development of alternative methods.

In our previous study, we discovered a strong correlation between urinary oxygen partial pressure and renal organ function impairment in children with sepsis. Building upon traditional biochemical indicators such as blood lactic acid levels, we will incorporate non-invasive tests like urine partial pressure of oxygen, renal ultrasound, and cardiac ultrasound, as well as novel markers like KIM-1, to establish a model for early recognition and assessment of kidney damage in children with sepsis. By utilizing commonly used biomarkers and the precise effects of urinary oxygen partial pressure, we aim to improve early identification and accurate intervention evaluation for pediatric sepsis kidney injury. This research will provide a crucial foundation for the development of early warning systems, diagnostic guidelines, and treatment protocols for pediatric sepsis kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* From May 2021 to December 2024, the study focused on patients admitted to the Pediatric Intensive Care Unit (PICU) for a duration exceeding three days. Specifically, patients with severe infection and those who underwent pediatric neurosurgery were diagnosed with sepsis according to the international standard for childhood sepsis established in 2005, the 2012 Surviving Sepsis Campaign guidelines for pediatric sepsis, and the 2015 expert consensus on sepsis criteria for Chinese children with septic shock. The age range of the patients included in the study spanned from 1 month to 16 years old.

Exclusion Criteria:

* Children who enter PICU 24 hours and die or exit PICU within 24 hours; Genetic metabolic diseases; Congenital immune deficiency; Can't sign an informed consent form.

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: Between the period of May 2021 to December 2024, the study focused on patients who were admitted to the Pediatric Intensive Care Unit (PICU) for a duration exceeding three days. Specifically, patients with a diagnosis of sepsis were selected based on the internationally recognized 2005 standard for childhood sepsis, the 2012 Surviving Sepsis Campaign guidelines for pediatric sepsis, and the 2015 expert consensus on sepsis criteria for Chinese children with septic shock. The age range of the patients included in the study spanned from 1 month to 16 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | the first three day after admission
  Alterations and specific biomarkers of the intestinal microbiota in patients with sepsis complicated by acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Yaya Xu, M.S., Study Director — Shanghai Jiaotong University School of Medicine Xinhua Hospital
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No